CLINICAL TRIAL: NCT06715540
Title: An Open-Label, Non-Comparative Study of the Safety, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of Ascending Doses of BCD-261 After Single Subcutaneous Injection in Healthy Subjects
Brief Title: Safety, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of Ascending Doses BCD-261 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BCD-261-1
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: anti-TL1A; anti-TNF-like ligand 1A; Ulcerative Colitis; Inflammatory Bowel Disease; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Intervention Model Description: Stage 1: "3+3" design (dose escalation). Stage 2: parallel arms (dose expansion)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1 (Experimental): Subjects in Cohort 1 will receive BCD-261 at a dose 1 during the Stage 1. Depending on the DLT, the cohort may include 1 to 3 subjects.
  Interventions: Drug: BCD-261, dose 1
- Cohort 2 (Experimental): Subjects in Cohort 2 will receive BCD-261 at a dose 2 during the Stage 1. Depending on the DLT, the cohort may include 3 to 6 subjects.
  Interventions: Drug: BCD-261, dose 2
- Cohort 3 (Experimental): Subjects in Cohort 3 will receive BCD-261 at a dose 3 during the Stage 1. Depending on the DLT, the cohort may include 3 to 6 subjects.
  Interventions: Drug: BCD-261, dose 3
- Cohort 4 (Experimental): Subjects in Cohort 4 will receive BCD-261 at a dose 4 during the Stage 1. Depending on the DLT, the cohort may include 3 to 6 subjects.
  Interventions: Drug: BCD-261, dose 4
- Cohort 5 (Experimental): Subjects in Cohort 5 will receive BCD-261 at a dose 5 during the Stage 1. Depending on the DLT, the cohort may include 3 to 6 subjects.
  Interventions: Drug: BCD-261, dose 5
- Cohort 6 (Experimental): Subjects in Cohort 6 will receive BCD-261 at a dose 6 during the Stage 1. Depending on the DLT, the cohort may include 3 to 6 subjects.
  Interventions: Drug: BCD-261, dose 6
- Cohort 7 (Experimental): Subjects in Cohort 7 will receive BCD-261 at a pre-specified proposed therapeautic dose X during the Stage 2. DLT events will not be assesed during the Stage 2.
  Cohort 7 will enroll 6 caucasian healthy subjects, who will recieve single subcutaneous injection of BCD-261 solution in vials.
  Interventions: Drug: BCD-261, pre-specified therapeautic dose X
- Cohort 8 (Experimental): Subjects in Cohort 8 will receive BCD-261 at a pre-specified proposed therapeautic dose X during the Stage 2. DLT events will not be assesed during the Stage 2.
  Cohort 8 will enroll 6 caucasian healthy subjects, who will recieve single subcutaneous injection of BCD-261 solution in pre-filled syringes.
  Interventions: Drug: BCD-261, pre-specified therapeautic dose X
- Cohort 9 (Experimental): Subjects in Cohort 9 will receive BCD-261 at a pre-specified proposed therapeautic dose X during the Stage 2. DLT events will not be assesed during the Stage 2.
  Cohort 9 will enroll about 10 asian healthy subjects, who will recieve single subcutaneous injection of BCD-261 solution in pre-filled syringes.
  Interventions: Drug: BCD-261, pre-specified therapeautic dose X
- Cohort 10 (Experimental): Subjects in Cohort 10 will receive BCD-261 at a pre-specified proposed therapeautic dose Y during the Stage 2. DLT events will not be assesed during the Stage 2.
  Cohort 10 will enroll about 10 asian healthy subjects, who will recieve single subcutaneous injection of BCD-261 solution in pre-filled syringes.
  Interventions: Drug: BCD-261, pre-specified therapeautic dose Y

INTERVENTIONS:
Drug: BCD-261, dose 1 — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in vials
  Other Names: anti-TL1A
  Arms: Cohort 1
Drug: BCD-261, dose 2 — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in vials
  Other Names: anti-TL1A
  Arms: Cohort 2
Drug: BCD-261, dose 3 — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in vials
  Other Names: anti-TL1A
  Arms: Cohort 3
Drug: BCD-261, dose 4 — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in vials
  Other Names: anti-TL1A
  Arms: Cohort 4
Drug: BCD-261, dose 5 — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in vials
  Other Names: anti-TL1A
  Arms: Cohort 5
Drug: BCD-261, dose 6 — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in vials
  Other Names: anti-TL1A
  Arms: Cohort 6
Drug: BCD-261, pre-specified therapeautic dose X — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in vials
  Other Names: anti-TL1A
  Arms: Cohort 7
Drug: BCD-261, pre-specified therapeautic dose X — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in pre-filled syringes
  Other Names: anti-TL1A
  Arms: Cohort 8; Cohort 9
Drug: BCD-261, pre-specified therapeautic dose Y — Anti-TL1A human monoclonal antibody. Solution for Subcutaneous Injection in pre-filled syringes
  Other Names: anti-TL1A
  Arms: Cohort 10

SUMMARY:
The goal of this clinical trial is to investigate the safety, tolerability, pharmacodynamics, pharmacokinetics, and immunogenicity of BCD-261 after single subcutaneous injection at ascending doses and proposed therapeutic doses to healthy male subjects aged from 18 to 45 years old.

The study consists of the first stage (dose escalation) and the second stage (dose expansion).

DETAILED DESCRIPTION:
The study is conducted in 2 stages. During the Stage 1 of the study, dose escalation is performed in several cohorts to assess the effects of dose-limiting toxicity (DLT), the maximum tolerated dose of BCD-261.

During the dose escalation one subject ("sentinel volunteer") will be included in cohort 1. Starting from the 2nd cohort and up to the 6th cohort, the study is planned within a classic "3+3" design.

Based on the results of the analysis of the Stage 1 data, including the assessment of safety, pharmacodynamics, pharmacokinetics, immunogenicity of BCD-261, a decision will be made on the possibility of switching to the Stage 2 of the study (dose expansion).

DLT events will be monitored for 7 days after BCD-261 injection (during Stage 1), and may include any of CTCAE 5.0 grade ≥3 adverse events that are at least possibly related to the study drug.

During the Stage 2 an extended study of the safety, pharmacodynamics, pharmacokinetics, and immunogenicity of BCD-261 at two pre-selected proposed therapeutic doses, is carried out with the inclusion of several additional cohorts of healthy caucasians and asians.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. For cohorts 1-8: Male subjects aged 18 to 45 years at the time of signing the ICF. For cohorts 9-10: Asian male subjects aged 18 to 45 years inclusive at the time of signing the ICF.
3. The ability of the subject to follow the Protocol procedures, in the Investigator's opinion.
4. A diagnosis of "healthy", established according to standard clinical, laboratory, and instrumental methods of examination carried out at screening, according to the assessment of the Investigator, as well as historical data (absence of acute and chronic diseases of the respiratory, cardiovascular, nervous systems, gastrointestinal tract, impaired liver or kidney function).
5. Hemodynamic parameters within the normal range: systolic blood pressure (SBP) ranging 100 to 130 mmHg, diastolic (DBP) ranging 60 to 90 mmHg, pulse ranging 60 to 90 bpm at screening.
6. Willingness of the subjects and their female partners of childbearing potential to use reliable contraceptive methods from the moment of signing the ICF, throughout the main study period, and up to Day 57 inclusive. This requirement does not apply to participants who have undergone surgical sterilization.
7. Willingness of subjects with reproductive potential to refrain from donating sperm, starting from the moment of signing the ICF, throughout the main study period until Day 57 inclusive.
8. Willingness to refrain from participating in any other clinical trials, starting from the moment of signing the ICF and throughout the study.
9. Willingness to refrain from vaccination with any vaccines during the period from the moment of signing the ICF until Day 127 of the study inclusive.

Exclusion Criteria:

1. Any medical or social condition that, in the opinion of the Investigator, prevents participation in this study.
2. Any confirmed or suspected immunosuppressive or immunodeficiency condition.
3. Any acute infectious and non-infectious diseases, including the period of convalescence, within 4 weeks from the moment of clinical recovery to signing the ICF, as well as during screening.
4. Diagnosis of infectious mononucleosis (documented or reported by the subject) within 2 months before signing the ICF and during screening.
5. Vaccination with live vaccines within 8 weeks and with any other vaccines within 4 weeks prior to signing the ICF and during screening.
6. A history of allergies and signs of other significant adverse reactions after the administration of any medicinal products.
7. Hypersensitivity to the components of BCD-261.
8. Body mass index (BMI) outside the normal range (18.0 to 30.0 kg/m2).
9. Results of standard laboratory and instrumental tests outside the normal ranges adopted at the study site.
10. Positive results of screening tests for HIV, hepatitis B and C, tuberculosis.
11. Repeated positive urine drug test, repeated positive saliva alcohol test at screening.
12. Impossibility of venipuncture for blood sampling (e.g., due to skin diseases at the sites of venipuncture).
13. Administration and use of the following drugs:

    * Regular oral or parenteral administration of any medicinal products, including over-the-counter drugs, vitamins, and dietary supplements, within less than 14 calendar days prior to estimated date of ID assignment.
    * A history of using anti-TL1A monoclonal antibodies.
    * Taking medications, including over-the-counter drugs, that have a pronounced effect on hemodynamics and liver function (barbiturates, omeprazole, cimetidine, etc.), within less than 30 days before the estimated date of ID assignment.
    * Taking drugs that affect the immune status (cytokines and their inducers, glucocorticoids, etc.) within less than 60 days before the estimated date of ID assignment.
14. Smoking of more than 10 cigarettes a day.
15. Consumption of more than 10 units of alcohol per week (1 unit of alcohol is equivalent to ½ L of beer, 200 mL of wine or 20 mL of spirits) or a history of alcoholism, drug addiction or drug abuse.
16. Surgical interventions performed less than within 90 days before the signing of the ICF.
17. Donation of 450 mL or more of blood or plasma within 60 days prior to signing the ICF.
18. Participation in any clinical study of medicinal products within 90 days before signing the ICF; previous participation in the same study with the exception of subjects who withdrew before the administration of the investigational product.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with adverse reactions | 127 days
Proportion of subjects with serious adverse reactions | 127 days
Proportion of subjects with CTCAE 5.0 grade 3 or higher adverse reactions | 127 days
Proportion of subjects who prematurely withdrew from the study due to adverse reactions | 127 days

OTHER OUTCOMES:
Cmax (Maximum concentration) | 127 days
Tmax (Time of maximum observed concentration) | 127 days
T1/2 (Elimination half-life period) | 127 days
Kel (Elimination rate constant) | 127 days
Cl (Clearance) | 127 days
Vd (Volume of distribution) | 127 days
Cmin (Minimum observed concentration) | 127 days
AUC(0-1344) (Area under curve from 0 to 1344 hours) | 57 days
AUC(0-inf) (Area under curve from 0 to infinity) | 127 days

CONTACTS AND LOCATIONS:
Overall Officials: Arina V Zinkina-Orikhan, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (1):
- "Meditsinskiy teсhnologiy Maly", Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Trials | BIOCAD — https://ct.biocad.ru/en/nozology?utm_source=biocad.ru&utm_medium=referral&utm_campaign=biocad_referral&utm_reffere=biocad.ru